CLINICAL TRIAL: NCT06969157
Title: Diagnosis and Its Procedural Pattern Among Patients Who Underwent Surgery at Aloha Medical Mission in Dhankuta, 2018
Acronym: Diagnosis and
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 3600
Record Dates: First submitted 2025-02-23; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Surgery With General Anesthesia
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgery — Minor or major surgeries were performed depending upon the primary diagnosis. Major surgery was defined as one done under general anesthesia while minor was one done under local anesthesia.

SUMMARY:
This was a retrospective, cross-sectional study of the Aloha medical mission in 2018, which involved analyzing recorded data on the sociodemographic profiles of patients, diseases, and surgical procedures. The data of patients was recorded using a pro forma, then entered into Excel and a coding list, and the data analysed using EZR.

ELIGIBILITY:
Inclusion Criteria:

* patients with complete records of age, gender, diagnosis, procedure performed, anesthesia type, perioperative complications and direct cost per patient.

Exclusion Criteria:

* patients with missing records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing surgery (major or minor) during the study period
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
frequency and distribution of surgical conditions | Through hospital stay, up to 7 days
  Type of surgery performed will be recorded based on operative notes and categorized by anatomical site and procedure type

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient information is available from corresponding author on reasonable request.
Supporting Information: SAP, ICF
Time Frame: It will be available infinitely after publication of the article.